CLINICAL TRIAL: NCT06441890
Title: BRE-10: BIomarker OptimizatioN of NeOadjuVAnt Therapy in BrEast Cancer: The INNOVATE Trial
Brief Title: BRE-10: Biomarker Optimization of Neoadjuvant Therapy in Breast Cancer
Acronym: BRE-10
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kent F. Hoskins, MD, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1384
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; 130-nm albumin-bound paclitaxel; Docetaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Treatment Arm (Other): One of the following Taxane options below per physician's choice
  * Paclitaxel 80mg/m2 IV D1, 8, 15 Q21 days
  * Nab-paclitaxel1 125mg/m2 IV D1, 8, 15 Q21 days
  * Docetaxel1 75mg/m2 IV D1 Q-21 days
  * Trastuzumab2 8mg/kg loading, then 6mg/kg IV/SQ D1 Q21 days
  * Pertuzumab2 840 mg loading, then 420mg IV/SQ D1 Q21 days
  * 1 may be substituted for paclitaxel for patients intolerant to paclitaxel or the steroid premed regimen, or at investigator discretion
  * 2 Pertuzumab, trastuzumab, and hyaluronidase injection for subcutaneous use may be substituted with dose per package insert
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Docetaxel; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Paclitaxel — 80mg/m2 IV D1, 8, 15
Drug: Nab-paclitaxel — 125mg/m2 IV D1, 8, 15
Drug: Docetaxel — 75mg/m2 IV D1
Drug: Trastuzumab — 8mg/kg loading, then 6mg/kg IV/SQ D1
Drug: Pertuzumab — 840 mg loading, then 420mg IV/SQ D1

SUMMARY:
Adult men and women with early-stage, IHC/FISH-defined HER2-positive breast cancer will have a MammaPrint®/BluePrint® assay performed on the diagnostic biopsy specimen, ordered by the treating Oncologist as standard care

DETAILED DESCRIPTION:
Adult men and women with early-stage, IHC/FISH-defined HER2-positive breast cancer will have a MammaPrint®/BluePrint® assay performed on the diagnostic biopsy specimen, ordered by the treating Oncologist as standard care. Patients whose tumors have a HER2-enriched molecular subtype on the MammaPrint®/BluePrint® assay and are recommended for neoadjuvant chemotherapy by their treating Oncologist will be recruited for study enrollment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at time of consent
* ECOG performance status 0, 1, or 2
* Histologically confirmed invasive breast cancer documented by core needle or surgical biopsy with 90 days prior to study registration.
* HER2-positive by IHC or FISH according to ASCO/CAP 2018 guidelines
* HER2-enriched subtype on the MammaPrint/BluePrint gene expression profile within 90 days prior to study registration.
* Curative resection of primary breast tumor(s) is planned; ipsilateral axillary nodes will be sampled by sentinel lymph node biopsy or axillary dissection
* Treating Oncologist recommends neoadjuvant chemotherapy
* No evidence of distant metastatic disease
* AJCC clinical stage: cT1c-T3, cN0-N2
* Baseline left ventricular ejection fraction (LVEF) of at least 50% on Echo or MUGA scan within 90 days prior to registration.

Adequate organ function as defined below:

Leukocytes ≥2,000/mm3 Platelet count ≥ 75,000/mm3 Absolute Neutrophil Count (ANC) ≥ 1,000/mm3 Hemoglobin (Hgb) ≥ 9.0 g/dL Creatinine/Calculated Creatine clearance (CrCI) Cr < 1.5 x upper limit of normal (ULN) or CrCl ≥ 50 mL/min using the Cockcroft-Gault formula Bilirubin ≤ 1.5 × ULN. Subjects with Gilbert's syndrome may have a bilirubin > 1.5 × ULN, if no evidence of biliary obstruction exists Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN

* Patients with synchronous bilateral primary breast tumors or multiple ipsilateral primary breast tumors are eligible if the treating Oncologist determines that the assigned treatment regimen is appropriate therapy for all primary tumors requiring chemotherapy.
* Able to provide written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization. or the Legally Authorized Representative (LAR) is able to provide consent and HIPAA authorization.
* Women of childbearing potential must agree to use a barrier form of contraception if they are sexually active with a male partner and cannot be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
* Patients with history of HIV/AIDS (acquired immunodeficiency syndrome) are eligible for this study if they are receiving anti-retroviral therapy and it does not include any medications known to alter metabolism or tolerability of component drugs in the protocol treatment regimen and the following criteria is met:

  - Patients without a history of AIDS-defining opportunistic infections within the past 12 months.
* Patients with Hepatitis B (HBV): chronic carriers of HBV infection (HBsAg-positive) or individuals who have serologic evidence of a resolved prior HBV infection (i.e., HBsAg-negative and anti-HBc-positive) are eligible if they are receiving appropriate suppressive antiviral therapy that does not include medications known to alter metabolism or tolerability of component drugs in the protocol treatment (see Appendix) prior to initiation of cancer therapy, and liver function tests meet study eligibility criteria.
* Patients with Hepatitis C (HCV): patients with a history of HCV infection who have completed curative antiviral treatment are eligible if the HCV RNA viral load is below the limit of quantification within 90 days of study enrollment. Patients on concurrent HCV treatment must have HCV RNA viral load below the limit of quantification within 30 days of study enrollment. Patients must also meet liver function test eligibility requirements and antiviral therapy does not include medications known to alter metabolism or tolerability of component drugs in the protocol treatment

Exclusion Criteria

* Any prior therapy for this breast cancer
* Active infection requiring systemic therapy at the time of study registration
* Pregnant or nursing
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Other major comorbidity (e.g., compromised liver function, major cardiovascular or cerebrovascular event within the past 6 months, uncontrolled diabetes mellitus or hypertension), as determined by treating physician.
* Any contraindication for any chemotherapy drug used in the assigned regimen.
* Baseline sensory neuropathy > grade 1
* History of hypersensitivity to any of the drugs in the treatment regimen. Patients with history of hypersensitivity may be treated on this protocol with either nab-paclitaxel or docetaxel.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have a pathological complete response (pCR) | 16 weeks
  This is defined as the absence of any residual invasive carcinoma on hematoxylin and eosin evaluation of the resected breast specimen and any resected lymph node tissue

SECONDARY OUTCOMES:
Participant outcomes using the Quality of Life (QOL) and EORTC QOL-C30 questionnaires | Baseline
  Number of participants having good outcome versus low outcomes. High score means worse health outcomes and low score means better health outcomes
Participant outcomes using the Quality of Life (QOL) and EORTC QOL-C30 questionnaires | 30 days post treatment
  Number of participants having good outcome versus low outcomes. High score means worse health outcomes and low score means better health outcomes
Participant outcomes using the Quality of Life (QOL) and EORTC QOL-C30 questionnaires | 6 months post treatment
  Number of participants having good outcome versus low outcomes. High score means worse health outcomes and low score means better health outcomes
Safety of the study treatment with be assessed by evaluating the number of participants experiencing Adverse Events (AEs) | 30 days post treatment
  AEs will be evaluated using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5
Treatment tolerability will be assessed | 30 days post treatment
  Number of participants that have cycle treatment delays
Treatment tolerability will be assessed | 30 days post treatment
  Number of participants that have cycle treatment cancelations
Treatment tolerability will be assessed | 30 days post treatment
  Number of participants that have dose reductions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Chicago, Illinois, United States